CLINICAL TRIAL: NCT04398836
Title: Preoperative Nutrition for Crohn's Disease Patients
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Director, R&D Department, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0825-18TLV
Record Dates: First submitted 2019-07-18; First posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Malnutrition; Crohn Disease
MeSH Terms: conditions — Malnutrition; Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Malnourished patients - EEN (Active Comparator): patiens will receive EEN for 4 week prior surgery
  Interventions: Dietary Supplement: Exclusive Enteral Nutrition
- Malnourished patients - enriched diet (Other): patiens will receive an enriched high energy and protein diet.
  Interventions: Other: High energy / protein diet.
- Well nourished patients (Other): Patient will receive a standard nutrition
  Interventions: Other: Standard nutrition

INTERVENTIONS:
Dietary Supplement: Exclusive Enteral Nutrition — Mulnourished patients will drink an enteral polymeric formula suited to their energy expenditure calculated by 25-30 kcal/kg and at least 1 gr/kg of protein, a minimum of 1500 ml (1500 kcal, 54 gr of protein). The amount of formula to achieve nutritional requirements are based on body weight, but the average intake is of 6-8 cups of formula (36-48 scoops of formula mixed with 1260-1680 ml of water to achieve a concentration of 1 kcal per ml). During this period patients will be guided to avoid eating and drinking anything but the enteral formula. The formula will be supplied to the patients by the investigators. The formula used for this study will be VITAL - suitable for people with disease-related malnutrition and malabsorption. Vital 1.5kcal is peptide-based, nutritionally complete formulation for the dietary management of active phase of Crohn's disease. VITAL includes all the nutritional macro and micronutrients and can serve as a sole source of nutrition.
  Arms: Malnourished patients - EEN
Other: High energy / protein diet. — Mulnourished patients will receive a high energy / protein diet.
  Arms: Malnourished patients - enriched diet
Other: Standard nutrition — Well nurished patients will receive a standard nutrition
  Arms: Well nourished patients

SUMMARY:
The investigator hypothesizes that compliance to Exclusive enteral nutrition (EEN) will be high among patients on an operation for their bowel disease, compared to the compliance rate seen in the general Crohn's Disease (CD) population.

Also,the investigator hypothesizes that clinical outcomes would improve, and post-operative complication rate will be reduces in malnourished CD patients receiving pre-operative 4 weeks EEN during the 4 weeks post-surgery, compared to CD patients receiving high energy and protein diet without EEN.

DETAILED DESCRIPTION:
Study design:

A randomized, none-blinded study. Study population: 144 CD patients designated for surgery, 96 malnourished patients and 44 well-nourished patients. Participants will be recruited from the Department of Gastroenterology, from Surgery Department and from the Nutrition Unit in the Tel Aviv Medical Center (TLVMC).

Study procedure CD patients who are awaiting surgery will be screened and randomly assigned to the study. After the decision to perform surgery and patient's acceptance to participate in the study but not more than 3 months before scheduled surgery, patient will undergo nutritional assessment. Patients suffering from malnutrition will be randomly assigned to the EEN group or to the group receiving enriched high energy and protein diet. Well-nourished patients will continue with standard nutritional therapy. Malnutrition will be defined according to Subjective Global Assessment (SGA)

Screening procedure:

Patients assigned to the interventional arm would be asked to adhere to EEN for two days prior to inclusion in order to assess tolerability and adherence to the assigned diet. Those who are not able to adhere to a two day EEN diet , will be withdrawn from the interventional arm, and will be treated with a high energy, high protein diet as the control group in accordance to the study protocol.

Study group:

Patients will drink an enteral polymeric formula suited to their energy expenditure calculated by 25-30 kcal/kg and at least 1 gr/kg of protein, a minimum of 1500 ml (1500 kcal, 54 gr of protein). The amount of formula to achieve nutritional requirements are based on body weight, but the average intake is of 6-8 cups of formula (36-48 scoops of formula mixed with 1260-1680 ml of water to achieve a concentration of 1 kcal per ml). During period patients guided to avoid eating and drinking anything but the enteral formula. The formula will be supplied to the patients by the investigators.

The formula used for this study will be VITAL - suitable for people with disease-related malnutrition and malabsorption. Vital 1.5kcal is peptide-based, nutritionally complete formulation for the dietary management of active phase of CD. VITAL includes all the nutritional macro and micronutrients and can serve as a sole source of nutrition. In cases of severe nutritional deterioration throughout the study, supplemental parenteral nutrition will be considered.

Control group:

Nutritional support by high energy/high protein diet, calculated by 25-30 kcal/kg and at least 1 gr/kg of protein. In cases of significant nutritional deterioration throughout the study, oral nutritional supplements or supplemental parenteral nutrition will be considered.

Well-nourished patient group: accepted standard nutritional therapy.

Compliance and dietary evaluation:

Patients will fill-up a 3 day food diary during every study visit to assesses recent dietary composition. Adherence to therapy will also monitored using the Medication Adherence Rating Scale (MARS) questionnaire.

Nutrients intake will be computed with the Israeli nutritional software "Zameret". Patients in the EEN group will be required to return the empty enteral formula containers.

Compliance to the diet instructed for the patient will be concidured as intake of 80% of calories per patient.

Compliance to the diet instructed for the patient will be concidured as intake of 80% of calories per patient.

Tolerability to EEN:

Tolerance will be defined as ingestion of the entire amount of formula requested by the patient without the development of any allergic/intolerant symptoms. Tolerance will be monitored during every study visit.

Disease activity:

Disease activity will be evaluated by serum C- Reactive Protein (CRP) concentration, fecal calprotectin concentration and Harvey-Bradshaw index (HBI).

Metabolic evaluation

Anthropometric measurements:

* Weight and height will be measured on a digital medical scale and body mass index (BMI) will be calculated.
* Handgrip strength will be measured by a handgrip dynamometer (JAMAR® - hydraulic hand dynamometer )
* Nutritional assessment by SGA questioners.
* Body composition by body electrical impedance.
* Resting Energy Expenditure (REE) will be measured by indirect calorimetry (Fitmate- Cosmed/ Italy)

Biochemical tests:

All blood samples will be drawn at the morning following 12 hours fast: albumin, blood count, serum CRP concentration and fecal calprotectin concentration.

Post operative clinical course:

Patient post-operative course will be documented from patients medical file. Parameters will include: hospitalization length, blood transfusions and other interventions, post operative medical treatment.

Fecal samples:

Stool will be analyzed for fecal calprotectin and for characterizing the microbial composition

Assessment of surgical complications

The following complications will be monitored 30d after surgery:

* Hospital readmissions
* Revision of surgery
* Stoma complications
* Severe bleeding
* Thrombotic event
* Ileus
* Liver complications
* Renal complications
* Infectious complications: Surgical site infection, Urinary tract infection, Pulmonary; anastomotic leaks, intraabdominal abscess and formation of new fistula.

Safety EEN is an accepted and recommended therapy for CD patients and considered a first-line therapy for inducing remission in children.

ELIGIBILITY:
Inclusion Criteria:

• CD patients awaiting surgery

Exclusion Criteria:

* Pregnancy and lactation
* Subjects on TPN
* Subjects with chronic conditions such as cancer, organ transplant subjects, advanced kidney or liver disease, systemic inflammatory conditions other than IBD
* Inability to sign informed consent and complete study protocol
* Surgical procedure to reverse ileostomy/colostomy or abscess drainage

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Compliance to diet | during every study visit week 0, week 1, week 2, week 3, week 4, 30 days post - surgery
  During every study visit compliance to diet instructed, monitor every week since initiating: week 0, week 4, 30 days post - surgery by 3 days food diary calculated average consumption of kcal and protein in grames.
  The same assessment carried out at week 1, week 2, week 3, by 24 - hour recall questionnaire.
  High Compliance considered if Calories > 80% protein ≥ 1 gr/kg from the expected metabolic assessment needs for each week 1-4 dietary intervention, and present better outcomes.
  1. using the MARS questionnaire - Medication Adherence Rating Scale. The patient should be asked to respond to the statements in the questionnaire by circling the answer which best describes their behaviour or attitude towards their medication during the past week.
  2. Patients will fill-up a 3 day food diary during every study visit to assesses recent dietary composition
Changes in adherence to therapy | during every study visit week 1, week 2, week 3, week 4, 30 days post - surgery
  During every study visit week 1, week 2, week 3, week 4, 30 days post - surgery, MARS, Medication Adherence Rating Scale - questionnaire filled by subject: Patient asked to respond to the statements in the questionnaire by circling the answer best describes their behavior or attitude towards their diet prescription during the past week. Score range between: min of 10-19 - no adherence to diet, 40-49 often adherence, 50 max score present permanent adherence.
Changes in tolerability to the diet | Tolerance will be monitored during every study visit: week 0, week 1, week 2, week 3, week 4
  Tolerance will be monitored during every study visit week 0, week 1, week 2, week 3, week 4, as ingestion of the entire amount of formula requested by the patient without the development of any allergic/intolerant symptoms, report on changes in tolerance documented and monitored in tailored form.

SECONDARY OUTCOMES:
The rate of post-operative complications in malnourished CD patients receiving pre-operative 4 weeks EEN, is changed during the 4 weeks post-surgery, compared to CD patients receiving high energy and protein diet without EEN one month after surgery. | One month after surgery
  Patient post-operative course documented from patients' medical file. Parameters include: hospitalization length, blood transfusions and other interventions, post - operative medical treatment and complications.

CONTACTS AND LOCATIONS:
Overall Officials: Nitsan Maharshak, MD, Principal Investigator — Tel Aviv Medical Center
Locations (1):
- Dep. of Gastroenterology, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No